CLINICAL TRIAL: NCT04788927
Title: Development of a Comprehensive Predictive Model for Risk of Metastatic Disease in PPGLs Based on a Combination of Clinical, Biochemical, Genetic, and Pathoanatomical Characteristics a Retrospective National Cohort Study
Brief Title: Development of a Predictive Model for the Risk of Metastatic Disease in PPGLs, a Retrospective Cohort Study
Acronym: PPGL-Pred
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor Ulla Feldt-Rasmussen, Rigshospitalet, Denmark
Other Study IDs: PPGL-Pred
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Paraganglioma; Pheochromocytoma; Genetic Predisposition to Disease; Pathology; Somatic Mutation; Head and Neck Cancer; Neuroendocrine Tumors
Keywords: Paraganglioma; Phaeochromocytoma; Clinical genetics; Pathology; Translational research
MeSH Terms: conditions — Paraganglioma; Pheochromocytoma; Genetic Predisposition to Disease; Head and Neck Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples and tumour tissue samples from existing biobanks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Phaeochromocytomas and paragangliomas (PPGLs) are tumours of the adrenal medulla and extra-adrenal sympathetic nervous system, some which can become metastatic. It is a very rare disease and the tumours are often detected late. Approximately 50 % of the tumours are caused by germline genetic variants screening programmes are recommended for patients and their family members; however, they are not yet well-targeted with respect to individual prognosis. In this study the investigatorscaim to characterize the genotype-phenotype associations in all Danish patients (n=400) diagnosed with PPGLs who have been followed in tertiary centres using medical records and national registries. To this end novel immunohistochemical, genetic, and epigenetic biomarkers in tumour tissues samples from biobank material (blood samples and tumour tissue) will be investigated to develop a comprehensive predictive algorithm for disease prognosis. The study will provide a clinical tool for an improved targeted screening program and subsequently prevention of disease development.

DETAILED DESCRIPTION:
Phaeochromocytomas and paragangliomas (PPGLs) are tumours of the adrenal medulla and extra-adrenal sympathetic nervous system, respectively, that often secrete catecholamines(1). The tumours are derived from the neural crest and approximately 50% are caused by a germline variant. Because of the strong heritability, genetic testing is recommended in all patients with PPGLs (2-5). Most PPGLs are non-malignant (defined as non-metastatic) tumours and respond well to surgical treatment. Approximately 15% of PPGLs are metastatic and incurable by currently available therapies(1). The latest WHO Blue Book classifies all PPGLs as possibly malignant due to their unpredictable behaviour(6).

PPGLs are very heterogeneous tumours predisposed by more than 20 distinct genes(1). In two thirds of the tumours a germline or somatic variant can be identified and thus PPGLs have been divided into distinct biological subgroups on the basis of these variants(1). A consensus statement from 2017 stated the necessity for a targeted gene panel (Next-Generation Sequencing, NGS) in all PPGL patients and testing of tumour DNA if possible to identify potential future targets for drug therapies(2). Furthermore, epigenetic changes in PPGLs and other endocrine tumours have been shown to be associated with the risk of metastatic disease(7-11) and future research should be focused on understanding both epigenetic and genetic changes in PPGLs as this will open opportunities for targeted molecular therapies and personalized medicine(11,12). It has been demonstrated that DNA methylation-based tumour classification is a valuable asset for clinical decision making(13).

Many histopathological predictive risk factors for poor prognosis have been proposed and scoring systems have been developed to identify those PPGLs that have a metastatic potential. The PASS (Pheochromocytoma of the Adrenal Gland Scaled Score) and GAPP (Grading system for Adrenal Phaeochromocytoma and Paraganglioma) scores are the most well-known (1,14-18). In a recent meta-analysis the algorithms were evaluated and it was concluded that both algorithms had a low positive predictive value but a high negative predictive value for PPGLs which indicated that the models were relevant for ruling out metastatic potential for both tumour types rather than identifying cases with an increased risk of disseminated disease. This could most probably be attributed to subjective assessment of criteria involved in these scoring systems. The authors concluded that the inclusion of NGS data and an overall molecular approach is needed to accurately pinpoint cases at risk for future metastases(19). Furthermore, there is a need for an algorithm based on objective measurements to ensure objectivity in the pathological diagnosis of PPGLs, similar to algorithms for adrenocortical carcinomas like the Helsinki Score and the Reticulin Algorithm(19-21). To this end computer-assisted techniques have shown promising results(11,20).

Correctly identifying PPGLs with a future risk of metastatic disease is a clinical challenge which impacts not only the physicians but also the patients and their family members. Today's clinical guidelines are based on 'rule all in' methods which have a costly impact on the healthcare resources and the quality of life of the patients. An algorithm based on histopathological, genetic, epigenetic, and clinical variables may be helpful in stratifying patients into risk categories with different needs for clinical follow-up.

Pilot Study: Patients followed at Copenhagen University Hospital, Copenhagen have been part of a pilot study on the effect of genetic screening of family members with SDHX variants on the clinical presentation of cases. Variants of the SDHX (SDHA, -AF2, -B, -C, -D) genes are a frequent cause of familial PPGLs. The investigators found distinct differences in the clinical and histopathological characteristics between genetic variants in SDHB. Family screening for SDHB variants resulted in earlier detection of tumours in two families. Patients with SDHA, SDHC and SDHD variants also had severe phaenotypes, underlining the necessity for a broad genetic screening of the proband. The study corroborated previous findings of poor prognostic markers and found that the genetic variants and clinical phenotype are linked and therefore useful in the decision of clinical follow-up. This study has been presented as master thesis at the University of Copenhagen 2019 (Grade A) and the manuscript has been published(22). The study corroborates the feasibility of the current project.

Process of the study

Part 1: Description of the genotype-phaenotype association in a nation-wide cohort of approximately 400 patients with PPGLs or germ-line genetic variants predisposing to PPGLs using clinical data, biochemical variables, tumour characteristics and imaging results. This national cohort will provide characterization of patients making it possible to identify a metastatic and non-metastatic clinical course, respectively.

Part 2: Identification of novel prognostic biomarkers using formalin-fixed paraffin-embedded tumor tissue samples for genetic testing (NGS for somatic variants), DNA methylation, PASS scoring, and immunohistochemical markers. Twenty patients with a poor prognosis (proof of metastases) and 20 patients with a good prognosis (non-metastatic) will be included from the Capital Region of Denmark. The results will be used to develop a new algorithm for clinical prognosis.

Part 3: Validation of the new algorithm in a second subcohort of patients with tumor tissue specimens selected at random from the national cohort. Tumor specimens will be subjected to investigation of the same novel prognostic biomarkers identified in part 2. Results will be entered into the new algorithm to test whether the clinical course can be accurately predicted.

Dissemination Positive, negative or inconclusive results will be published in peer-reviewed international journals and presented at scientific meetings and in relevant patient fora. The study group members are affiliated to ENDO-ERN (European Reference Network on Rare Endocrine Conditions), a European collaboration of highly specialized centres treating rare endocrine conditions through which results can be disseminated (https://endo-ern.eu/).

To ensure completeness and transparency in the reporting of results the investigators will use the STROBE reporting guidelines relevant to cohort studies.

Patient involvement:

Patients with lived experiences contribute additional expertise and give valuable, novel insights and thus improve the effectiveness of the study. Furthermore, the patient perspective is essential in the presentation of the results. Relevant patients with the disease in question from our outpatient clinic will be invited to participate in the Steering Committee.

Safety and ethical considerations Treatment of personal data: General Data Protection Regulation will be strictly adhered to. Approval by the Ethics Committee for the Capital Region has been granted (H-20065699, 19th of February 2021).

Database: The database will be established under RedCap, which is accessible nation-wide and managed centrally by the data protection unit of The Capital Region.

Statistics: Based on previous studies which have developed similar algorithms (20,21) the investigators will need approximately 200 patients to achieve statistical power in relation to validation of the algorithm in the larger cohort. Study population characteristics will be presented using descriptive statistics. Group differences will be tested primarily using non-parametric tests (Mann-Whitney, Wilcoxon) or t-test. Associations between the genotype and phaenotype will be analysed by ANOVA (analysis of variance) and regression analysis controlling for relevant confounders, i.e. age and sex, where appropriate. The sensitivity and specificity of the algorithm to predict poor or good outcome will be determined using multiple regression analyses, Chi2 and ROC (Receiver Operating Characteristics). The investigators will seek help from professional statisticians at Copenhagen University at Statistical Advisory Service for PhD-students and students at the Faculty of Health Sciences.

ELIGIBILITY:
Inclusion Criteria:

* All Danish patients diagnosed with PPGLs or genetic variants that predispose to PPGLs since 1996 will be included.

Exclusion Criteria:

* None from the initial data collection. If there are no tumour tissue or blood samples from a patient in the biobanks they will subsequently be excluded.

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Location: Nation-wide cohort of all patients followed in one of the tertiary hospitals: Copenhagen (Rigshospitalet), Århus (Skejby) and Odense University hospital.
  Identification: The patients will be retrieved from the National Danish Registry of Hospital Diagnoses by use of their national identification number (CPR).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Malignant or non-malignant disease | 25 ys (1996-2021) retrospective data collection of approximately 400 patients until death or until today.
  Defined as metastatic disease

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Prof., Dr. med., Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - National University Hospital, Department of Medical Endocrinology, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicolas M, Dahia P. Predictors of outcome in phaeochromocytomas and paragangliomas. F1000Res. 2017 Dec 21;6:2160. doi: 10.12688/f1000research.12419.1. eCollection 2017. PMID 29333259
- [Background] NGS in PPGL (NGSnPPGL) Study Group; Toledo RA, Burnichon N, Cascon A, Benn DE, Bayley JP, Welander J, Tops CM, Firth H, Dwight T, Ercolino T, Mannelli M, Opocher G, Clifton-Bligh R, Gimm O, Maher ER, Robledo M, Gimenez-Roqueplo AP, Dahia PL. Consensus Statement on next-generation-sequencing-based diagnostic testing of hereditary phaeochromocytomas and paragangliomas. Nat Rev Endocrinol. 2017 Apr;13(4):233-247. doi: 10.1038/nrendo.2016.185. Epub 2016 Nov 18. PMID 27857127
- [Background] Pacak K, Tella SH. Pheochromocytoma and Paraganglioma. In: De Groot LJ, Chrousos G, Dungan K, et al., eds. Endotext. South Dartmouth MA: MDText.com, Inc.; 2000
- [Background] Plouin PF, Amar L, Dekkers OM, Fassnacht M, Gimenez-Roqueplo AP, Lenders JW, Lussey-Lepoutre C, Steichen O; Guideline Working Group. European Society of Endocrinology Clinical Practice Guideline for long-term follow-up of patients operated on for a phaeochromocytoma or a paraganglioma. Eur J Endocrinol. 2016 May;174(5):G1-G10. doi: 10.1530/EJE-16-0033. PMID 27048283
- [Background] Lenders JW, Duh QY, Eisenhofer G, Gimenez-Roqueplo AP, Grebe SK, Murad MH, Naruse M, Pacak K, Young WF Jr; Endocrine Society. Pheochromocytoma and paraganglioma: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2014 Jun;99(6):1915-42. doi: 10.1210/jc.2014-1498. PMID 24893135
- [Background] Lloyd RV OR, Klöppel G, Rosai J. WHO Classification of Tumours of Endocrine Organs 4th ed. Lyon IARC; 2017
- [Background] Oishi T, Iino K, Okawa Y, Kakizawa K, Matsunari S, Yamashita M, Taniguchi T, Maekawa M, Suda T, Oki Y. DNA methylation analysis in malignant pheochromocytoma and paraganglioma. J Clin Transl Endocrinol. 2016 Dec 23;7:12-20. doi: 10.1016/j.jcte.2016.12.004. eCollection 2017 Mar. PMID 29067245
- [Background] Lee SE, Oh E, Lee B, Kim YJ, Oh DY, Jung K, Choi JS, Kim J, Kim SJ, Yang JW, An J, Oh YL, Choi YL. Phenylethanolamine N-methyltransferase downregulation is associated with malignant pheochromocytoma/paraganglioma. Oncotarget. 2016 Apr 26;7(17):24141-53. doi: 10.18632/oncotarget.8234. PMID 27007161
- [Background] Backman S, Maharjan R, Falk-Delgado A, Crona J, Cupisti K, Stalberg P, Hellman P, Bjorklund P. Global DNA Methylation Analysis Identifies Two Discrete clusters of Pheochromocytoma with Distinct Genomic and Genetic Alterations. Sci Rep. 2017 Mar 22;7:44943. doi: 10.1038/srep44943. PMID 28327598
- [Background] Jouinot A, Assie G, Libe R, Fassnacht M, Papathomas T, Barreau O, de la Villeon B, Faillot S, Hamzaoui N, Neou M, Perlemoine K, Rene-Corail F, Rodriguez S, Sibony M, Tissier F, Dousset B, Sbiera S, Ronchi C, Kroiss M, Korpershoek E, de Krijger R, Waldmann J, K D, Bartsch, Quinkler M, Haissaguerre M, Tabarin A, Chabre O, Sturm N, Luconi M, Mantero F, Mannelli M, Cohen R, Kerlan V, Touraine P, Barrande G, Groussin L, Bertagna X, Baudin E, Amar L, Beuschlein F, Clauser E, Coste J, Bertherat J. DNA Methylation Is an Independent Prognostic Marker of Survival in Adrenocortical Cancer. J Clin Endocrinol Metab. 2017 Mar 1;102(3):923-932. doi: 10.1210/jc.2016-3205. PMID 27967600
- [Background] Jouinot A, Bertherat J. MANAGEMENT OF ENDOCRINE DISEASE: Adrenocortical carcinoma: differentiating the good from the poor prognosis tumors. Eur J Endocrinol. 2018 May;178(5):R215-R230. doi: 10.1530/EJE-18-0027. Epub 2018 Feb 23. PMID 29475877
- [Background] Pang Y, Liu Y, Pacak K, Yang C. Pheochromocytomas and Paragangliomas: From Genetic Diversity to Targeted Therapies. Cancers (Basel). 2019 Mar 28;11(4):436. doi: 10.3390/cancers11040436. PMID 30925729
- [Background] Capper D, Jones DTW, Sill M, Hovestadt V, Schrimpf D, Sturm D, Koelsche C, Sahm F, Chavez L, Reuss DE, Kratz A, Wefers AK, Huang K, Pajtler KW, Schweizer L, Stichel D, Olar A, Engel NW, Lindenberg K, Harter PN, Braczynski AK, Plate KH, Dohmen H, Garvalov BK, Coras R, Holsken A, Hewer E, Bewerunge-Hudler M, Schick M, Fischer R, Beschorner R, Schittenhelm J, Staszewski O, Wani K, Varlet P, Pages M, Temming P, Lohmann D, Selt F, Witt H, Milde T, Witt O, Aronica E, Giangaspero F, Rushing E, Scheurlen W, Geisenberger C, Rodriguez FJ, Becker A, Preusser M, Haberler C, Bjerkvig R, Cryan J, Farrell M, Deckert M, Hench J, Frank S, Serrano J, Kannan K, Tsirigos A, Bruck W, Hofer S, Brehmer S, Seiz-Rosenhagen M, Hanggi D, Hans V, Rozsnoki S, Hansford JR, Kohlhof P, Kristensen BW, Lechner M, Lopes B, Mawrin C, Ketter R, Kulozik A, Khatib Z, Heppner F, Koch A, Jouvet A, Keohane C, Muhleisen H, Mueller W, Pohl U, Prinz M, Benner A, Zapatka M, Gottardo NG, Driever PH, Kramm CM, Muller HL, Rutkowski S, von Hoff K, Fruhwald MC, Gnekow A, Fleischhack G, Tippelt S, Calaminus G, Monoranu CM, Perry A, Jones C, Jacques TS, Radlwimmer B, Gessi M, Pietsch T, Schramm J, Schackert G, Westphal M, Reifenberger G, Wesseling P, Weller M, Collins VP, Blumcke I, Bendszus M, Debus J, Huang A, Jabado N, Northcott PA, Paulus W, Gajjar A, Robinson GW, Taylor MD, Jaunmuktane Z, Ryzhova M, Platten M, Unterberg A, Wick W, Karajannis MA, Mittelbronn M, Acker T, Hartmann C, Aldape K, Schuller U, Buslei R, Lichter P, Kool M, Herold-Mende C, Ellison DW, Hasselblatt M, Snuderl M, Brandner S, Korshunov A, von Deimling A, Pfister SM. DNA methylation-based classification of central nervous system tumours. Nature. 2018 Mar 22;555(7697):469-474. doi: 10.1038/nature26000. Epub 2018 Mar 14. PMID 29539639
- [Background] Kulkarni MM, Khandeparkar SG, Deshmukh SD, Karekar RR, Gaopande VL, Joshi AR, Kesari MV, Shelke RR. Risk Stratification in Paragangliomas with PASS (Pheochromocytoma of the Adrenal Gland Scaled Score) and Immunohistochemical Markers. J Clin Diagn Res. 2016 Sep;10(9):EC01-EC04. doi: 10.7860/JCDR/2016/20565.8419. Epub 2016 Sep 1. PMID 27790441
- [Background] Bialas M, Okon K, Dyduch G, Ciesielska-Milian K, Buziak M, Hubalewska-Dydejczyk A, Sobrinho-Simoes M. Neuroendocrine markers and sustentacular cell count in benign and malignant pheochromocytomas - a comparative study. Pol J Pathol. 2013 Jun;64(2):129-35. doi: 10.5114/pjp.2013.36004. PMID 23900871
- [Background] Stenman A, Zedenius J, Juhlin CC. The Value of Histological Algorithms to Predict the Malignancy Potential of Pheochromocytomas and Abdominal Paragangliomas-A Meta-Analysis and Systematic Review of the Literature. Cancers (Basel). 2019 Feb 15;11(2):225. doi: 10.3390/cancers11020225. PMID 30769931
- [Background] Pennanen M, Heiskanen I, Sane T, Remes S, Mustonen H, Haglund C, Arola J. Helsinki score-a novel model for prediction of metastases in adrenocortical carcinomas. Hum Pathol. 2015 Mar;46(3):404-10. doi: 10.1016/j.humpath.2014.11.015. Epub 2014 Dec 9. PMID 25582500
- [Background] Duregon E, Fassina A, Volante M, Nesi G, Santi R, Gatti G, Cappellesso R, Dalino Ciaramella P, Ventura L, Gambacorta M, Dei Tos AP, Loli P, Mannelli M, Mantero F, Berruti A, Terzolo M, Papotti M. The reticulin algorithm for adrenocortical tumor diagnosis: a multicentric validation study on 245 unpublished cases. Am J Surg Pathol. 2013 Sep;37(9):1433-40. doi: 10.1097/PAS.0b013e31828d387b. PMID 23774167
- [Background] Main AM, Rossing M, Borgwardt L, Gronkaer Toft B, Rasmussen AK, Feldt-Rasmussen U. Genotype-phenotype associations in PPGLs in 59 patients with variants in SDHX genes. Endocr Connect. 2020 Aug;9(8):793-803. doi: 10.1530/EC-20-0279. PMID 32688340
- [Background] Ebbehoj A, Jacobsen SF, Trolle C, Robaczyk MG, Rasmussen AK, Feldt-Rasmussen U, Thomsen RW, Poulsen PL, Stochholm K, Sondergaard E. Pheochromocytoma in Denmark during 1977-2016: validating diagnosis codes and creating a national cohort using patterns of health registrations. Clin Epidemiol. 2018 Jun 13;10:683-695. doi: 10.2147/CLEP.S163065. eCollection 2018. PMID 29942158